CLINICAL TRIAL: NCT06522958
Title: Comparative Study of the Effects of Novel High Dissolving Transitional Foods on Post-Operative Outcomes for Patients Undergoing Craniofacial Surgery
Brief Title: Effect of Novel High Dissolving Transitional Foods
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-00648
Record Dates: First submitted 2024-07-23; First posted 2024-07-26 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Craniofacial Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients randomized to the intervention group will receive a high dissolving transitional food product.
  Interventions: Dietary Supplement: High Dissolving Transitional Food
- Standard of Care Group (No Intervention): Patients randomized to the standard of care group will not receive a high dissolving transitional food product.

INTERVENTIONS:
Dietary Supplement: High Dissolving Transitional Food — Transitional foods are solid foods that rapidly change texture in the presence of moisture (e.g., water or saliva) or temperature change. Duration of consumption of the investigational agent will include the time of the surgery until the second post-operative evaluation. This is estimated to be approximately 1-2 months in total.
  Arms: Intervention Group

SUMMARY:
This is a prospective comparative study, where patients who meet inclusion criteria undergoing a craniofacial procedure will either be provided with novel high dissolving transitional foods for use in the post-operative period (Intervention Group) or will not be provided the food and will proceed as per current standard of care (Standard of Care Group). Both groups will be followed pre-operatively at time of pre-operative visit, and will be followed in the post-operative period, with two visits at 1 and 3 weeks post-operatively, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 0 years, 6 months to 18 years of age
* Patients with a diagnosed cleft/craniofacial condition undergoing one of the following cleft/craniofacial related surgeries in the upcoming calendar year (a-c):

  1. Cleft Palate Repair (Palatoplasty)
  2. Alveolar Bone Graft Surgery
  3. Velopharyngeal Insufficiency Surgery
* Patients who eat fully by mouth (PO)
* Patients who adhered to scheduling protocols and attended all necessary pre- and post-operative visits

Exclusion Criteria:

* Patients under the age of 6 months or over the age of 18
* Patients who utilize an NG-tube or G-tube for primary means of nutrition/hydration
* Patients who have PO recommendations from a licensed Speech-Language Pathologist that prevents their ability to consume Level 4 IDDSI (pureed) foods, including patients who are NPO.
* Patients with any diagnosed allergies to the ingredients listed on the Savorease Therapeutic Foods ingredient labels
* Patients/caregivers who are not able to participate in pre- and post-operative protocoled visits for any reason
* Patients/caregivers who are not able to respond to written questions presented in English

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Caregiver-Reported Rating of Feeding Experience | Week 1 Post-Operation (Post-Op)
  Caregivers of participants will complete short survey to assess patient's feeding-related quality of life (QOL) related to the post-operative period. The survey comprises 10 items; each item utilizes a 5-point Likert scale ranging from 0 (Strongly Disagree) to 4 (Strongly Agree). The total score is the sum of responses and ranges from 0-40; lower scores indicate greater feeding-related QOL.
Caregiver-Reported Rating of Feeding Experience | Week 3 Post-Op
  Caregivers of participants will complete short survey to assess patient's feeding-related quality of life (QOL) related to the post-operative period. The survey comprises 10 items; each item utilizes a 5-point Likert scale ranging from 0 (Strongly Disagree) to 4 (Strongly Agree). The total score is the sum of responses and ranges from 0-40; lower scores indicate greater feeding-related QOL.

SECONDARY OUTCOMES:
Number of Participants with Wound Issues at Pre-Op Visit | Baseline (Pre-Op Visit)
  Participants will undergo a wound examination to assess for the presence of fistula, dehiscence, or wound complications.
Number of Participants with Wound Issues at Week 1 Post-Op | Week 1 Post-Op
  Participants will undergo a wound examination to assess for the presence of fistula, dehiscence, or wound complications.
Number of Participants with Wound Issues at Week 3 Post-Op | Week 3 Post-Op
  Participants will undergo a wound examination to assess for the presence of fistula, dehiscence, or wound complications.
30-Day Readmission Rate | Day 30 Post-Op
  Percentage of participants who are readmitted to the hospital within 30 days post-operation.
Average Participant Weight at Pre-Op Visit | Baseline (Pre-Op Visit)
  Participant weight is measured in pounds (lbs).
Average Participant Weight at Week 1 Post-Op | Week 1 Post-Op
  Participant weight is measured in pounds (lbs).
Average Participant Weight at Week 3 Post-Op | Week 3 Post-Op
  Participant weight is measured in pounds (lbs).
Number of Participants who Self-Report Use of Pain Medicine at Pre-Op Visit | Baseline (Pre-Op Visit)
Number of Participants who Self-Reported Use of Pain Medicine at Week 1 Post-Op | Week 1 Post-Op
Number of Participants who Self-Reported Use of Pain Medicine at Week 3 Post-Op | Week 3 Post-Op

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Flores, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Margaret.lico@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Margaret.lico@nyulangone.org . To gain access, data requestors will need to sign a data access agreement.